CLINICAL TRIAL: NCT00323674
Title: Prospective Randomized Study to Evaluate the Recovery of a Hernia Inguinalis by a Minimally Invasive Open Preperitoneal Surgery With Polysoft Mesh Versus a Classic Open Surgery According to Modified Lichtenstein Procedure With Light Weight Mesh
Brief Title: Minimally Invasive Open Preperitoneal Surgery With Polysoft Mesh Versus a Classic Open Surgery With Light Weight Mesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006/080
Record Dates: First submitted 2006-05-07; First posted 2006-05-09 (Estimated); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Hernia, Inguinal
Keywords: Hernia Inguinalis
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Light Weight Mesh (Active Comparator)
  Interventions: Device: Light Weight Mesh
- Polysoft Mesh (Active Comparator)
  Interventions: Device: Polysoft Mesh

INTERVENTIONS:
Device: Polysoft Mesh — Polysoft Mesh is used.
  Arms: Polysoft Mesh
Device: Light Weight Mesh — Light Weight Mesh is used.
  Arms: Light Weight Mesh

SUMMARY:
This is a prospective randomized study to evaluate the recovery of a hernia inguinalis by a minimally invasive open preperitoneal surgery with polysoft mesh versus a classic open surgery according to modified Lichtenstein procedure with light weight mesh.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic hernia inguinalis
* > 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2006-03 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08-31 (Actual)

PRIMARY OUTCOMES:
Percentage of relapse | Evaluation at day 0, 3 weeks, 3 months, 1 year and 3 year.
Postoperative pain assessment | Evaluation at day 0, 3 weeks, 3 months, 1 year and 3 year.
Duration to full recovery (able to do all activities) | Evaluation at day 0, 3 weeks, 3 months, 1 year and 3 year.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be